CLINICAL TRIAL: NCT04744493
Title: A Clinical Trial for Evaluation of the Safety and Effect of MR-guided FUS Subthalamotomy for Medication-refractory Parkinson's Disease Motor Features
Brief Title: A Clinical Trial for the Safety and Effect of MRGuided FUS Subthalamotomy for Medication Refractory Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PD003J
Record Dates: First submitted 2020-09-23; First posted 2021-02-09 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2020-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: This is a prospective, open-label, single-center, and sponsor-initiated clinical trial. The clinical trial follows the Clinical Investigation Plan, GCP.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm of Exablate 4000 as a single arm (Experimental): Only one arm of treatment by Exablate 4000 was established.
  Interventions: Device: ExaBlate 4000

INTERVENTIONS:
Device: ExaBlate 4000 — The Exablate 4000, an advanced, non-invasive technique for performing ablation of the Thalamus for treating Essential Tremor, received FDA PMA (P150038) approval for unilateral treatment of Essential Tremor in 2016.

SUMMARY:
Study design: This is a prospective, open-label, single-center, and sponsor-initiated clinical trial. The clinical trial follows the Clinical Investigation Plan, GCP. Objective: The objective of the clinical trial is to evaluate improving Parkinson's disease motor features by MR-guided focused ultrasound surgery (Patient who has less effectiveness.).

DETAILED DESCRIPTION:
Endpoint: All PD003J treated subjects will be followed up for 4 months. The primary endpoints will be safety of unilateral, PD003J subthalamotomy for PD. The endpoint will be determined from adverse events recorded during the 4 months period for safety. Secondary endpoints will include changes in MDS-UPDRS, levodopa equivalent medication, Global Impression of Change and so on.

Primary endpoint of safety: Incidence and severity of adverse events (AE/AEs) associated with PD003J treatment of idiopathic PD at 4 months post treatment. Safety will be evaluated individually for each subject who is treated. An analysis of safety will be performed on all treated subjects and will be determined by an evaluation of the incidence and severity of device- and procedure-related complications. In particular, in this study, the incidence of severe involuntary movements (one-sided ballism) is confirmed. All AEs will be reported and categorized by investigators as definitely, probably, possibly, unlikely, or unrelated to the device, subthalamotomy procedure, and/or Parkinson's disease progression.

Secondary endpoints: Secondary endpoints will include both comparison of baseline to 1 week visit, 2-month visit and baseline to 4-month visit assessments for the following: • MDS-UPDRS parts I, II, III, and IV • Levodopa equivalent medication usage (milligrams) • Patient and Physician Global Impression of Change • Patient Satisfaction Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, age 30 years and older
2. Subjects who are able and willing to give informed consent and able to attend all study visits through 4 Months
3. Subjects with a diagnosis of Parkinson's Disease using the MDS criteria as confirmed by a movement disorder neurologist at the site
4. Predominant disability from one side of the body (i.e. unilateral or markedly asymmetric disease) as determined by a movement disorders neurologist
5. Subjects should be on a stable dose of all PD medications for 30 days prior to study entry.
6. Topographic coordinates of the subthalamic nucleus are localizable on MRI so that it can be targeted by the PD003J.
7. Subject is able to communicate sensations during the PD003J procedure.
8. Subject cannot obtain with drugs for treating Parkinson's disease.

Exclusion Criteria:

1. Hoehn and Yahr stage in the ON medication state of 2.5 or greater
2. Presence of severe dyskinesia as noted by a score of 3 or 4 on questions 4.1 and 4.2 of the MDS-UPDRS
3. Presence of other central neurodegenerative disease suspected on neurological examination. These include: multisystem atrophy, progressive supranuclear palsy, corticobasal syndrome, dementia with Lewy bodies, and Alzheimer's disease.
4. Any suspicion that Parkinsonian symptoms are a side effect from neuroleptic medications
5. Subjects who have had deep brain stimulation or a prior stereotactic ablation of the basal ganglia
6. Presence of significant cognitive impairment defined as score ≤ 21 on the Montreal Cognitive Assessment (MoCA)
7. Unstable psychiatric disease, defined as active uncontrolled depressive symptoms, psychosis, delusions, hallucinations, or suicidal ideation. Subjects with stable, chronic anxiety or depressive disorders may be included provided their medications have been stable for at least 60 days prior to study entry and if deemed appropriately managed
8. Subjects with significant depression as determined following a comprehensive assessment. Significant depression is being defined quantitatively as a score of greater than 19 on the Beck Depression Inventory.
9. Subjects exhibiting any behavior(s) consistent with ethanol or substance abuse as defined by the criteria outlined in the DSM-IV as manifested by one (or more) of the following occurring within the preceding 12-month period:

   * Recurrent substance use resulting in a failure to fulfill major role obligations at work, school, or home (such as repeated absences or poor work performance related to substance use; substance-related absences, suspensions, or expulsions from school; or neglect of children or household).
   * Recurrent substance use in situations in which it is physically hazardous (such as driving an automobile or operating a machine when impaired by substance use)
   * Recurrent substance-related legal problems (such as arrests for substance related disorderly conduct)
   * Continued substance use despite having persistent or recurrent social or interpersonal problems caused or exacerbated by the effects of the substance (for example, arguments with spouse about consequences of intoxication and physical fights).
10. Subjects with unstable cardiac status including:

    * Unstable angina pectoris on medication
    * Subjects with documented myocardial infarction within six months of protocol entry
    * Significant congestive heart failure defined with ejection fraction < 40
    * Subjects with unstable ventricular arrhythmias
    * Subjects with atrial arrhythmias that are not rate-controlled
11. Severe hypertension (diastolic BP > 100 on medication)
12. History of or current medical condition resulting in abnormal bleeding and/or coagulopathy
13. Receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk or hemorrhage (e.g. Avastin) within one month of focused ultrasound procedure. For anticoagulants with washout period shorter than one week the minimum period of time between stopping this medication and ExAblate procedure will be in accordance with washout time as per official effective medication labeling.
14. Subjects with risk factors for intraoperative or postoperative bleeding as indicated by: platelet count less than 100,000 per cubic millimeter, a documented clinical coagulopathy, or INR coagulation studies exceeding the institution's laboratory standard
15. Patient with severely impaired renal function with estimated glomerular filtration rate <30mL/min/1.73m2 (or per local standards should that be more restrictive) and/or who is on dialysis;
16. Subjects with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.
17. Significant claustrophobia that cannot be managed with mild medication.
18. Subject who weigh more than the upper weight limit of the MR table and who cannot fit into the MR scanner
19. Subjects who are not able or willing to tolerate the required prolonged stationary supine position during treatment.
20. History of intracranial hemorrhage
21. History of multiple strokes, or a stroke within past 6 months
22. Subjects with a history of seizures within the past year
23. Subjects with malignant brain tumors
24. Subjects with lower limbarterial blood flow disorder
25. Subjects with intracranial aneurysms requiring treatment or arterial venous malformations (AVMs) requiring treatment.
26. Any illness that in the investigator's opinion preclude participation in this study.
27. Subjects unable to communicate with the investigator and staff.
28. Subject is pregnant or lactating
29. Subjects who is enrolled or will be enrolled in clinical study or clinical research
30. Subjects who have an Overall Skull Density Ratio of 0.30 or less as calculated from the screening CT

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence and severity of adverse events (AE/AEs) associated with PD003J treatment of idiopathic PD from baseline until 4 months post treatment. | Comfirmation from baseline until 4 months post treatment
  The primary safety outcome including incidence and severity of adverse events (AE/AEs) will be assessed at 4 months. The severity of any adverse events that will be reported by patients or that will be observed during the procedure or at 4 months post treatment will be assessed. A complication or worsening of a preexisting clinical condition after the procedure will be considered to be an adverse event regardless of causality.

SECONDARY OUTCOMES:
Secondary endpoints will include MDS-UPDRS parts I, II, III, and IV at baseline, 1 week, 2 months, and 4 months post treatment. | Comparison between baseline, 1 week, 2 months, and 4 months post treatment.
  The main efficacy assessment selects MDS-UPDRS Part I, II, III, and IV III of 11 items related to tremor and movement symptom variability, and difference in score from baseline before surgery to postoperative score. The degree of improvements of 11 items will be evaluated. The primary efficacy outcome will be the difference in the change from baseline to 4 months in the MDS-UPDRS motor score for the more affected body side in the off-medication state. The unabbreviated scale title, the minimum and maximum values, and whether higher scores mean a better or worse outcome will not be established for reporting outcome as efficacy.
Levodopa equivalent medication usage (milligrams). | Comparison between baseline, 1 week, 2 months, and 4 months post treatment.
  The following secondary data at baseline, 1 week, 2 months, and 4 months post treatment will be summarized using descriptive statistics and graphical methods:
  • Levodopa equivalent medication usage (milligrams) The unabbreviated scale title, the minimum and maximum values, and whether higher scores mean a better or worse outcome will not be established for reporting outcome as efficacy.
Patient and clinician Global Impression Rating Scale. | Comparison between baseline, 1 week, 2 months, and 4 months post treatment.
  The CGIC rating is made on a 7-point Likert-type scale where change from baseline is rated as marked improvement (1), moderate improvement (2), minimal improvement (3), no change (4), minimal worsening (5), moderate worsening (6), and marked worsening (7). The phisicians will evaluate the change between baseline and 3 evaluation points after treatment. The unabbreviated scale title, the minimum and maximum values, and whether higher scores mean a better or worse outcome will not be established for reporting outcome as efficacy.
Patient Satisfaction Questionnaire. | Comparison between baseline, 1 week, 2 months, and 4 months post treatment.
  The phisicians will evaluate the change between baseline and 3 evaluation points after treatment.The unabbreviated scale title, the minimum and maximum values, and whether Higher scores mean a better or worse outcome will not be established for reporting outcome as efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Osaka University Hospital, Suita, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No